CLINICAL TRIAL: NCT03530878
Title: Periacetabular Osteotomy Versus Arthroscopic Management of Mild Hip Dysplasia: A Randomized Clinical Trial
Brief Title: Mild Hip Dysplasia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rafael J. Sierra, M.D., Professor of Orthopedics, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-007229
Record Dates: First submitted 2018-04-09; First posted 2018-05-21 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Hip Dysplasia
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Arthroscopy (HA) (Experimental): This approach addresses intraarticular pathology in the form of labral tears and cartilage that are often concomitant with DDH 3. Furthermore, capsular plication can be performed through HA to reduce instability of the joint.
  Interventions: Procedure: Hip Arthroscopy
- Periacetabular Osteootmy (PAO) (No Intervention): The Bernese periacetabular osteotomy (PAO) remains the gold standard for treatment of symptomatic developmental dysplasia of the hip (DDH) in most patients with closed triradiate cartilage. First developed by Ganz in 1984, this technique utilizes 4 osteotomies to completely mobilize the acetabular fragment 1. Although a technically demanding procedure, it allows optimal correction in all planes and maintains integrity of the posterior column, enabling early weight bearing and mobilization.

INTERVENTIONS:
Procedure: Hip Arthroscopy — Intraarticular pathology in the form of labral tears and cartilage that are often concomitant with DDH
  Arms: Hip Arthroscopy (HA)

SUMMARY:
Hip dysplasia is a complex problem that exists on a spectrum from mild to severe disease. Periacetabular osteotomy (PAO) remains the gold standard for most patients with dysplasia; however, the procedure is quite invasive making the decision to proceed in cases of mild disease difficult. Hip arthroscopy (HA) is an alternative minimally invasive technique that can be used to address mild dysplasia. Nevertheless, HA has less capability for correction and in rare instances can exacerbate instability in the dysplastic hip. There is a paucity of data examining outcomes between these two treatment strategies for this challenging problem.

DETAILED DESCRIPTION:
The Bernese periacetabular osteotomy (PAO) remains the gold standard for treatment of symptomatic developmental dysplasia of the hip (DDH) in most patients with closed triradiate cartilage. First developed by Ganz in 1984, this technique utilizes 4 osteotomies to completely mobilize the acetabular fragment 1. Although a technically demanding procedure, it allows optimal correction in all planes and maintains integrity of the posterior column, enabling early weight bearing and mobilization. Several groups have confirmed the long-term efficacy of this joint preservation procedure with a recent report from the inventing institution documented impressive survivorship up to 30 years after surgery 2. Treatment with PAO is more controversial for mild forms of dysplasia where the lateral center-edge angle (LCEA) is 18° - 25° and/or the Tӧnnis angle is 8° - 15°. In these patients the delta correction is more limited, thus creating a more unpredictable result with equally invasive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of symptomatic mild DDH
* Lateral center-edge angle 18° - 25° and/or Tӧnnis angle 8° - 15°
* Skeletally mature
* Age 18 - 45
* Tonnis Grade 0 or 1 osteoarthritis (minimal or no arthritis)
* Ability to receive a standard of care preoperative MRI arthrogram of the hip

Exclusion Criteria:

* Pregnant women
* Neurogenic dysplasia
* Legg-Calvé-Perthes disease
* Previous surgery about the hip including previous hip arthroscopy to address intra-articular pathology

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
The Forgotten Joint Score-12 (FJS-12) | 1 year
  Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Rafael J Sierra, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials